CLINICAL TRIAL: NCT01815320
Title: A PILOT, EXPLORATIVE STUDY TO IDENTIFY CONTRAST-ENHANCED ULTRASOUND (CE-US) PATTERNS THAT CHARACTERIZE ACUTE ALLOGRAFT REJECTION AND OTHER CAUSES OF ACUTE ALLOGRAFT DYSFUNCTION IN RENAL TRANSPLANT RECIPIENTS
Brief Title: CE-US in Renal Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CE-US; 2010-019126-13 (EudraCT Number)
Record Dates: First submitted 2013-02-25; First posted 2013-03-21 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Renal Transplantation
Keywords: Renal Transplant; Contrast-enhanced ultrasound; Acute allograft rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast-enhanced ultrasound (CE-US) (Experimental): Ce-US is performed by contrast agent infusion SonoVue. The acquisition protocol will consist of two different administrations of SonoVue, performed 10 minutes apart. In the first session, SonoVue microbubbles will be administered as a fast 1.5 ml bolus immediately followed by 5 ml saline solution. In the second session, max 2 vials (9.6 ml) of SonoVue will be infused at an infusion rate between 0.5 and 1.0 ml/min.
  Interventions: Procedure: Contrast-enhanced ultrasound (CE-US); Device: SonoVue

INTERVENTIONS:
Procedure: Contrast-enhanced ultrasound (CE-US)
Device: SonoVue

SUMMARY:
Acute allograft dysfunction is often observed in the first weeks after kidney transplantation. Renal biopsy is universally considered the gold standard procedure for differential diagnosis of acute allograft dysfunction secondary to intraparenchymal causes. Kidney biopsy, however, is an invasive procedure that is time and cost consuming. Moreover, it may but not contribute to clinical diagnosis in about 10% of cases because of the impossibility to perform the analysis or of inadequacy of the biopsy sample. Availability or readily applicable non-invasive procedures might therefore allow increasing the performance of differential diagnosis of allograft dysfunction. In the recent years, a novel US imaging technique, namely contrast-enhanced ultrasound (CE-US),has been developed. The agent used in this study, Sonovue microbubbles consist of a central sulphur hexafluoride core with a surrounding phospholipid monolayer and last for several minutes in the systemic circulation before spontaneous degradation with absorption of the gaseous component by the lungs and the phospholipid shell by the liver. With the use of gasfilled microbubbles that act as scatterers within the blood stream and the development of low-MI ultrasound techniques that allow the visualization of the bubbles without destroying them, it is possible to improve the depiction of vessels and have access to structural and functional information on the microcirculation. Moreover SonoVue microbubbles are not nephrotoxic and can be safely used to evaluate kidney disfunction.

Thus, whether a. different patterns of parenchymal perfusion detected by CE-US can be associated with different patterns of renal graft involvement during acute renal function deterioration and b. whether, conversely, different patterns of parenchymal perfusion detected by CE-US may help predicting different patterns of renal involvement will be investigated in 20 deceased or living donor kidney graft recipients.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Kidney transplantation with a functioning graft (dialysis independence)
* Clinical indication to histologic evaluation of the kidney graft
* Written Informed consent (according to the Declaration of Helsinki guidelines)

Exclusion criteria:

* Specific contraindications to histologic evaluation of the kidney graft (bleeding time > 15 min, intra-abdominal implantation of the graft)
* Known hypersensitivity to sulphur hexafluoride or to any of the components of SonoVue.
* Recent Acute Coronary Syndrome (ACS) or clinically unstable ischaemic cardiac disease, including: evolving or ongoing myocardial infarction, typical angina at rest within last 7 days, significant worsening of cardiac symptoms within last 7 days, recent coronar artery intervention or other factors suggesting clinical instability (for example, recent deterioration of ECG, laboratory or clinical findings), acute cardiac failure, Class III/IV cardiac failure, or severe rhythm disorders.
* Right-to-left shunts, severe pulmonary hypertension (PAP >90 mmHg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Changes in complete or partial occlusion of pre-glomerular arteries and arterioles;changes in functional (and reversible) vasoconstriction of pre-glomerular arteries and arterioles. | At week 1,2,3 and 4.
  All examinations will be done by Contrast-enhanced ultrasound. Contrast agent wash-in (sec) and contrast agent wash-out (sec) will be assessed.
Changes in interstitial edema and cellular infiltration with tubulitis; changes in interstitial edema with tubular cell necrosis. | At week 1,2,3 and 4.
  All examinations will be done by Contrast-enhanced ultrasound. Contrast agent wash-in (sec) and contrast agent wash-out (sec) will be assessed.
Changes in complete or partial occlusion of pre-glomerular arteries and arterioles; changes in functional (and reversible) vasoconstriction of pre-glomerular arteries and arterioles. | At month 2,3,4,5,6,7,8,9,10,11,and 12.
  All examinations will be done by Contrast-enhanced ultrasound. Contrast agent wash-in (sec) and contrast agent wash-out (sec) will be assessed.
Changes in interstitial edema and cellular infiltration with tubulitis; changes in interstitial edema with tubular cell necrosis. | At month 2,3,4,5,6,7,8,9,10,11,and 12.
  All examinations will be done by Contrast-enhanced ultrasound. Contrast agent wash-in (sec) and contrast agent wash-out (sec) will be assessed.

SECONDARY OUTCOMES:
Changes in CE-US parameters from episodes of acute allograft deterioration versus baseline | At the time of acute allograft episode, assessed up to 12 months.
  All examinations will be done by Contrast-enhanced ultrasound. Contrast agent wash-in (sec) and contrast agent wash-out (sec) will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Unità di Nefrologia e Dialisi - A.O. Papa Giovanni XXIII, Bergamo, Bergamo, Italy